CLINICAL TRIAL: NCT01688323
Title: Identification of Predictors of Tolerance to Chemoradiotherapy in Elderly Patients With Head and Neck Cancer
Brief Title: Finding Predictors of Side Effects to Chemoradiation Treatment in Elderly Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1208; 12-0805 (Other: UNC IRB)
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Head and Neck Cancer
Keywords: Geriatrics; Oncology; Biological Markers; Survey Instruments; p16; Geriatric Oncology; Biological Markers of Aging; Symptom Assessment; Cancer; Older Persons; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Surveys and Questionnaires; Geriatric Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elderly Chemorads: Elderly patients with Head and Neck Cancer who are Undergoing Chemotherapy
  Interventions: Other: Collect Blood and Survey Instruments

INTERVENTIONS:
Other: Collect Blood and Survey Instruments — Each subject will be administered the appropriate surveys and blood draws over the course of the study.
  Other Names: Geriatric Assessment; FACT-HN; p16 Expression; Health Behavior Questionnaire

SUMMARY:
To look at what types of measures can be used to predict how an older person will tolerate chemoradiation treatment for head and neck cancer. This study uses surveys and a blood draw to look at the different measures.

DETAILED DESCRIPTION:
Purpose: To identify baseline predictors of change in function over the course of treatment with chemoradiotherapy in patients with head and neck cancer.

Participants: Patients 65 or older who have an appointment at the North Carolina Cancer Hospital (NCCH) or other participating sites, have planned chemoradiotherapy for head and neck cancer

Procedures (methods): Consenting subjects will complete a Geriatric Assessment, Functional Assessment of Cancer Therapy - Head and Neck and give a blood sample for CBC and p16INK4a at the start of their chemoradiotherapy, at week four, at the end and 90 days post therapy. They will also complete a health behavior questionnaire at baseline.

ELIGIBILITY:
Inclusion Criteria

* Patients will be eligible for this protocol provided they have an appointment at the North Carolina Cancer Hospital (NCCH), have planned chemoradiotherapy for head and neck cancer (any histology) and consent to complete the Geriatric Assessment. No exclusions will be made based on gender, ethnicity, performance status or race. Patient must be able to read and speak English.
* Signed, IRB approved written informed consent.
* Age of at least 65 years.
* Enrollment in other studies, both therapeutic and observational, will not result in exclusion.

Exclusion Criteria

* Inability to read and speak English.
* Inability to comply with study for any other reason than language

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly (65 and older) patients with Head and Neck Cancer
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Significant Change in Function from Baseline to Post-Treatment | 2 years
  To determine if there is a significant change in the Instrumental Activities of Daily Living (IADL) subscore of the Geriatric Assessment (GA) from baseline to 90 days post-treatment.

SECONDARY OUTCOMES:
Explore Association between Baseline Measures and Decline in Living Status | 2 years
  To explore the association of baseline measures with time to decline in living status. (For example, completely independent to requiring home help, or requiring home help to moving to a nursing home, etc.)
Explore Association of Baseline Measures with Grade 3 or Higher Toxicity | 2 years
  To explore the association of baseline measures with the occurrence of any grade 3 or higher toxicity as a consequence of chemoradiotherapy.
Explore Association of Baseline p16 with Baseline GA Measures | 2 years
  To explore the association of baseline p16 expression with baseline subscores of the Geriatric Assessment.
Explore Changes in p16 Expression, GA Subscales and FACT-HN Scores Over Time. | 2 years
  To explore changes in p16 expression, GA subscales, and FACT-HN scores over the course of treatment
Explore Association between Baseline Measures and Changes in IADL Subscore | 2 years
  To explore the association of baseline measures with change in IADL subscore.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Geriatric Oncology Program — https://unclineberger.org/patientcare/programs/geriatric